CLINICAL TRIAL: NCT04543409
Title: A Multicenter, Randomized, Double-blind, Parallel-group, Placebo Controlled Study to Investigate the Use of Benralizumab for Eosinophilic Esophagitis
Brief Title: A Study of Benralizumab in Patients With Eosinophilic Esophagitis
Acronym: MESSINA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: High-level results from the MESSINA Phase III trial showed that AstraZeneca's Fasenra (benralizumab) did not meet one of the two dual-primary endpoints. Given the lack of clear benefit in this patient population, study has been terminated.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D3255C00001; 2019-002871-32 (EudraCT Number)
Record Dates: First submitted 2020-08-18; First posted 2020-09-10 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-10

CONDITIONS: Eosinophilic Esophagitis
Keywords: Eosinophilic Esophagitis; EoE; Benralizumab
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — benralizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Benralizumab (Experimental): Benralizumab active solution will be administered SC to patients by healthcare professionals in this clinical study using an accessorized prefilled syringe (APFS)
  Interventions: Biological: Benralizumab
- Placebo (Placebo Comparator): Placebo solution will be administered SC to patients by healthcare professionals in this clinical study using an accessorized prefilled syringe (APFS)
  Interventions: Biological: Matching placebo

INTERVENTIONS:
Biological: Benralizumab — Solution for injection in a single accessorized prefilled syringe (APFS) will be administered subcutaneously (SC), 1 mL fill volume
  Arms: Benralizumab
Biological: Matching placebo — Matching placebo solution for injection in APFS, 1 mL fill volume. Placebo solution will be administered subcutaneously (SC), 1 mL fill volume
  Arms: Placebo

SUMMARY:
The aim of this Phase 3 study is to investigate the use of benralizumab as a treatment for patients with EoE. The effect of doses of benralizumab on EoE histologic signs and symptoms will be assessed over a 52-week treatment period (including a 24-week double-blind placebo-controlled treatment period and a 28-week open-label treatment period). It is proposed that benralizumab will deplete eosinophils from GI tissue(s), improve the symptoms of dysphagia, and improve endoscopy scores as well as other markers of disease activity. Upon completion of the initial 52-week treatment period, patients will be offered an additional Open Label Extension period of at least 1 year, with benralizumab treatment and ongoing study assessments.

ELIGIBILITY:
Inclusion Criteria:

* Patients 12 to 65 years of age, inclusive, at the time of signing the informed consent or assent (if applicable) form.
* Documented previous diagnosis of EoE by endoscopy.
* Must be symptomatic at Visit 1 (screening) and Visit 2 (randomization):

  1. A patient reported an average of at least 2 days per week with an episode of dysphagia over the 4 weeks prior to Visit 1 AND
  2. An average of at least 2 days per week with an episode of dysphagia (Daily DSQ ≥2) between Visit 1 and Visit 2, and at least 2 days per week with an episode of dysphagia (Daily DSQ ≥2) in each of the 2 weeks immediately prior to randomization
* May be on background medications for EoE and related treatments during the study as long as the background medications have been stable for at least 4 weeks (8 weeks for PPI) prior to the screening and there is agreement not to change type of background medication or dosage during the run-in period and for the first 52 weeks of the study unless a change is medically indicated.
* Negative serum pregnancy test for female patients of childbearing potential at Visit1.
* Women of childbearing potential must agree to use a highly effective form of birth control (confirmed by the Investigator) from randomization throughout the study duration and within 12 weeks after last dose if IP.

Exclusion Criteria:

* Other GI disorders such as active Helicobacter pylori infection, history of achalasia, esophageal varices, Crohn's disease, ulcerative colitis, inflammatory bowel disease, or celiac disease.
* Esophageal stricture that prevents the easy passage of a standard endoscope or any critical esophageal stricture that requires dilation during the run-in period.
* Esophageal dilation performed within 8 weeks prior to screening and prior esophageal surgery that would impact the assessments for EoE
* Use of a feeding tube, or having a pattern of not eating solid food daily during the run-in period.
* Hypereosinophilic syndrome, defined by multiple organ involvement and persistent blood eosinophil count >1500 eos/μL.
* EGPA vasculitis.
* Eosinophilic gastritis, gastroenteritis, enteritis, or colitis documented by biopsy.
* Current malignancy, or history of malignancy with some specific exceptions.
* History of anaphylaxis to any biologic therapy or vaccine.
* Current active liver disease:

  * Chronic stable hepatitis B and C (including positive testing for hepatitis B surface antigen [HBsAg] or hepatitis C antibody), or other stable chronic liver disease are acceptable if patient otherwise meets eligibility criteria.
  * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level ≥3 times the upper limit of normal (ULN), confirmed by repeated testing during the run-in period.
* Helminth parasitic infection diagnosed within 24 weeks prior to the date informed consent or assent (if applicable) is obtained that has not been treated with or has failed to respond to standard of care therapy.
* History of known immunodeficiency disorder including a positive human immunodeficiency virus (HIV) test.
* Concomitant use of immunosuppressive medication.
* Initiation or change of a food-elimination diet regimen or reintroduction of a previously eliminated food group in the 6 weeks prior to start of the run-in period.
* Currently pregnant, breastfeeding, or lactating women.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2022-09-19 (Actual); Study Completion 2023-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc E. Rothenberg, MD, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (68):
- United States (20):
  - Research Site, Little Rock, Arkansas
  - Research Site, St. Petersburg, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Normal, Illinois
  - Research Site, Park Ridge, Illinois
  - Research Site, White Marsh, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Chesterfield, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, Lincoln, Nebraska
  - Research Site, Ocean City, New Jersey
  - Research Site, New York, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Uniontown, Pennsylvania
  - Research Site, Salt Lake City, Utah
  - Research Site, Richmond, Virginia
- Canada (4):
  - Research Site, Hamilton, Ontario
  - Research Site, London, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Windsor, Ontario
- France (6):
  - Research Site, Dijon
  - Research Site, Lille
  - Research Site, Lyon
  - Research Site, Pessac
  - Research Site, Suresnes
  - Research Site, Toulouse
- Germany (3):
  - Research Site, Frankfurt
  - Research Site, München
  - Research Site, Remscheid
- Israel (5):
  - Research Site, Afula
  - Research Site, Holon
  - Research Site, Kfar Saba
  - Research Site, Petah Tikva
  - Research Site, Tel Aviv
- Italy (6):
  - Research Site, Florence
  - Research Site, Genova
  - Research Site, Napoli
  - Research Site, Pisa
  - Research Site, Rozzano
  - Research Site, Verona
- Japan (4):
  - Research Site, Chiba
  - Research Site, Izumo-shi
  - Research Site, Maebashi
  - Research Site, Osaka
- Netherlands (3):
  - Research Site, Amsterdam
  - Research Site, Nieuwegein
  - Research Site, Nijmegen
- Poland (8):
  - Research Site, Gdansk
  - Research Site, Knurów
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Rzeszów
  - Research Site, Szczecin
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Russia (2):
  - Research Site, Chelyabinsk
  - Research Site, Moscow
- Spain (4):
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, Bilbao
  - Research Site, Madrid
- United Kingdom (3):
  - Research Site, Brighton
  - Research Site, Darlington
  - Research Site, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Rothenberg ME, Dellon ES, Collins MH, Bredenoord AJ, Hirano I, Peterson KA, Brooks L, Caldwell JM, Fjallbrant H, Grindebacke H, Ho CN, Keith M, McCrae C, Sinibaldi D, White WI, Datto CJ; MESSINA Trial Investigators. Eosinophil Depletion with Benralizumab for Eosinophilic Esophagitis. N Engl J Med. 2024 Jun 27;390(24):2252-2263. doi: 10.1056/NEJMoa2313318. PMID 38924732
- See also: This is a poster. — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3255C00001&attachmentIdentifier=ac52d6ea-ef76-4f2a-80d2-34c1df605954&fileName=947_Messina_US_Poster_(Interactive)_V2.0_Master.pdf&versionIdentifier=
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3255C00001&attachmentIdentifier=c3793f8e-7115-402a-865c-0f76c155a81d&fileName=D3225C00001_-_CSR_Synopsis_Redacted.pdf&versionIdentifier=
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3255C00001&attachmentIdentifier=d160d7cd-a701-4e6b-8a07-8ef644b8ec45&fileName=D3255C00001_MESSINA_CSP_v_7.0_2022-04-01_Redacted.pdf&versionIdentifier=
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3255C00001&attachmentIdentifier=87647f3b-e786-4778-a814-2f15b19693fe&fileName=D3255C00001_SAP_v4_Final_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 404 participants were screened between 22SEP2020 and 22FEB2022. Of those, 211 were randomized to either the treatment (104 participants) or placebo (107 participants) arms of the double-blind treatment period. One participant, who did not meet inclusion/exclusion criteria, was incorrectly randomized but not dosed. Therefore, 103 participants started in the treatment arm and 107 in the placebo arm, for a total of 210 participants.
Pre-assignment Details: All patients completed a run-in period of 2 to 8 weeks during which inclusion/exclusion criteria was assessed, medical history taken, endoscopy with biopsies performed, and patient reported outcomes (PROs), clinical laboratories, and diet questionnaires were administered.
Groups:
- Benralizumab: 30mg Benralizumab injection delivered subcutaneously every 4 weeks
- Placebo: Matching Placebo injection delivered subcutaneously every 4 weeks through week 24, then 30mg Benralizumab injection delivered subcutaneously every 4 weeks after week 24
Period: Double-Blind Treatment Period
Arm/Group | Benralizumab | Placebo
Started | 103 | 107
Completed | 101 | 106
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Subject perceives the IP to be ineffective. | 1 | 0
Period: Open-Label Treatment Period
Arm/Group | Benralizumab | Placebo
Started | 100 (One participant enrolled in OL treatment period off study drug (not included in this count).) | 105 (One participant chose not to enroll in the OL treatment period.)
Completed | 79 | 82
Not Completed | 21 | 23
Not completed — Lost to Follow-up | 0 | 1
Not completed — Study terminated by sponsor | 17 | 19
Not completed — Withdrawal by Subject | 4 | 3
Period: Open-Label Extension Treatment Period
Arm/Group | Benralizumab | Placebo
Started | 45 (34 participants from previous period chose not to enroll in optional OLE period.) | 48 (34 participants from previous period chose not to enroll in optional OLE period.)
Completed | 0 | 0
Not Completed | 45 | 48
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Study terminated by sponsor | 44 | 44
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Unable to schedule gastroscopy | 0 | 1
Not completed — No study/treatment discontinuation information | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who were randomized and received any IP were included in the full analysis set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Benralizumab | Placebo | Total
Number analyzed (Participants) | 103 | 107 | 210
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.9 (13.49) | 33.6 (12.73) | 33.7 (13.08)
Age, Customized [Number; unit: Participants] — Age Group 1
  Participants
    < 18 years old | 14 | 14 | 28
    18-21 years old | 11 | 11 | 22
    22-35 years old | 32 | 35 | 67
    >= 36 years old | 46 | 47 | 93
Age, Customized [Number; unit: Participants] — Age Group 3
  Participants
    <= 21 years old | 25 | 25 | 50
    > 21 years old | 78 | 82 | 160
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 22 | 53
  Male | 72 | 85 | 157
Race/Ethnicity, Customized [Number; unit: Participants] — Population: Race and ethnicity are missing for all French participants due to local regulation rules.
  Participants
    Black or African American: number analyzed (Participants) | 103 | 104 | 207
    Black or African American | 1 | 1 | 2
    White: number analyzed (Participants) | 103 | 104 | 207
    White | 97 | 96 | 193
    Native Hawaiian or other Pacific Islander: number analyzed (Participants) | 103 | 104 | 207
    Native Hawaiian or other Pacific Islander | 0 | 1 | 1
    American Indian or Alaska Native: number analyzed (Participants) | 103 | 104 | 207
    American Indian or Alaska Native | 0 | 0 | 0
    Asian: number analyzed (Participants) | 103 | 104 | 207
    Asian | 2 | 5 | 7
    Other: number analyzed (Participants) | 103 | 104 | 207
    Other | 3 | 1 | 4
Race/Ethnicity, Customized [Number; unit: Participants] — Ethnicity Group Population: Race and ethnicity are missing for all French participants due to local regulation rules.
  Participants
    Hispanic or Latino: number analyzed (Participants) | 103 | 104 | 207
    Hispanic or Latino | 6 | 10 | 16
    Non-Hispanic or Latino: number analyzed (Participants) | 103 | 104 | 207
    Non-Hispanic or Latino | 97 | 94 | 191

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With a Histologic Response, Defined as a Peak Esophageal Intraepithelial Eosinophil Count ≤ 6 Eos/Hpf.
Description: Percentage of patients with a histologic response at Week 24 and Week 52. A histologic response is defined as a peak esophageal intraepithelial eosinophil count <= 6 eos/hpf across all available esophageal levels. Subjects with no biopsy data at Week 24 or with intercurrent events prior to Week 24 such as changes to background medications or additional new therapies for EoE are considered non-responders.
  The number analyzed represents the number of participants in the treatment group that could have made it to the timepoint by the data cut off.
Time Frame: Week 24, Week 52
Population: Full analysis set (All randomized participants who received at least one dose of IP).
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 103 | 107
Percentage of Participants
  Week 24 | 87.4 [80.97 to 93.79] | 6.5 [1.86 to 11.23]
  Week 52: number analyzed (Participants) | 46 | 47
  Week 52 | 82.6 [71.66 to 93.56] | 89.4 [80.55 to 98.18]
Statistical Analysis 1: Comparison: Benralizumab vs Placebo; Analysis completed at Week 24; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 117.49, 95% CI 2-sided [38.17 to 361.64] — The OR estimate and p-value was obtained from the CMH test controlling for region (North America and Rest of the world), baseline steroid use, and presence of strictures at baseline. Odds ratio values >1 favor Benra 30 mg treatment group

2. Primary Outcome: Changes From Baseline in Dysphagia Symptom Questionnaire (DSQ)
Description: The Dysphagia Symptom Questionnaire (DSQ) captures the presence and severity of dysphagia symptoms in the past day in a 4-item questionnaire. The DSQ score is calculated over 14-day periods and ranges from 0 to 84, with a lower score indicating less severe dysphagia. At least 8 days with evaluable daily score in 14-day period are required; otherwise the DSQ score for the period is set to missing.
  The number analyzed represents the number of participants with data at that visit (including patients with imputed values post intercurrent events).
Time Frame: Week 24, Week 52
Population: Full analysis set (All randomized participants who received at least one dose of IP).
Measure: Least Squares Mean (95% Confidence Interval); unit: Score
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 103 | 107
Score
  Week 24: number analyzed (Participants) | 95 | 100
  Week 24 | -12.102 [-16.05 to -8.15] | -15.101 [-19.02 to -11.19]
  Week 52: number analyzed (Participants) | 41 | 45
  Week 52 | -19.409 [-25.65 to -13.17] | -19.806 [-25.70 to -13.91]
Statistical Analysis 1: Comparison: Benralizumab vs Placebo; Analysis completed at Week 24; Test type: Superiority — For any patients with intercurrent events, the DSQ scores after the occurrence of those events were imputed using return-to-baseline MI. Missing data not due to intercurrent events were imputed using MI (MAR). Analysis was repeated on 100 imputed datasets, and results were combined using Rubin's formula; p = 0.1770, ANCOVA; Model: Change from baseline in DSQ = Treatment + baseline DSQ + Region + Baseline steroid use + Presence of strictures at baseline; Difference in Least Squares Means = 2.999, 95% CI 2-sided [-1.36 to 7.35]

3. Secondary Outcome: Percent Change From Baseline in Tissue Eosinophils
Description: Percent change from baseline in tissue eosinophils (eos) at Week 24 and Week 52.
  The number analyzed represents the number of participants with data at that visit (including imputed values).
Time Frame: Week 24, Week 52
Population: Full analysis set (All randomized participants who received at least one dose of IP).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of change
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 103 | 107
Percentage of change
  Week 24: number analyzed (Participants) | 97 | 100
  Week 24 | -94.8 [-100.00 to -82.45] | 1.4 [-11.75 to 14.60]
  Week 52: number analyzed (Participants) | 46 | 47
  Week 52 | -85.0 [-100.00 to -62.50] | -88.6 [-100.00 to -73.67]
Statistical Analysis 1: Comparison: Benralizumab vs Placebo; Analysis completed at Week 24; Test type: Superiority — For any patients with intercurrent events, the Peak Esophageal intraepithelial eosinophil (eos) counts after the occurrence of those events were imputed using return-to-baseline MI. Missing data not due to intercurrent events were imputed using MI (MAR); p < 0.0001, ANCOVA; Model: Percent change from baseline in Peak Esophageal intraepithelial eos counts = Treatment + baseline Peak Esophageal intraepithelial eos counts; Difference in Least Squares Means = -96.2, 95% CI 2-sided [-114.53 to -77.85]

4. Secondary Outcome: Change From Baseline in Eosinophilic Esophagitis-Histology Scoring System (EoE-HSS) Total Grade Score at Week 24
Description: EoE-HSS Grade and Stage Scores evaluate eight features: eosinophil density, basal zone hyperplasia, eosinophil abscesses, eosinophil surface layering, dilated intercellular spaces, surface epithelial alteration, dyskeratotic epithelial cells, and lamina propria fibrosis. Severity (grade) and extent (stage) of abnormalities will be scored using a 4-point scale (0 normal; 3 maximum change). Total grade score (TGS): mean of the grade score ratios per region. Grade score ratio per region is the sum of all available feature grade scores divided by the maximum possible score. The maximum possible total grade score is 1.
  The number analyzed represents the number of participants with data at that visit (including imputed values).
Time Frame: Week 24
Population: Full analysis set (All randomized participants who received at least one dose of IP).
Measure: Least Squares Mean (95% Confidence Interval); unit: Grade Score Ratio Change
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 97 | 100
Grade Score Ratio Change | -0.264 [-0.297 to -0.232] | -0.089 [-0.122 to -0.056]
Statistical Analysis 1: Comparison: Benralizumab vs Placebo; Test type: Superiority — For any patients with intercurrent events, the EoE-HSS total grade score after the occurrence of those events were imputed using return-to-baseline MI. Missing data not due to intercurrent events were imputed using MI (MAR); p < 0.0001, ANCOVA; Change from baseline in EoE-HSS TGS = Treatment + baseline EoE-HSS grade score + Region + Baseline steroid use + Presence of strictures at baseline; Difference in Least Squares Means = -0.175, 95% CI 2-sided [-0.21 to -0.14]

5. Secondary Outcome: Change From Baseline in Eosinophilic Esophagitis-Histology Scoring System (EoE-HSS) Total Stage Score at Week 24
Description: EoE-HSS Grade and Stage Scores evaluate eight features: eosinophil density, basal zone hyperplasia, eosinophil abscesses, eosinophil surface layering, dilated intercellular spaces, surface epithelial alteration, dyskeratotic epithelial cells, and lamina propria fibrosis. Severity (grade) and extent (stage) of abnormalities will be scored using a 4-point scale (0 normal; 3 maximum change). Total stage score (TSS): mean of the stage score ratios per region. Stage score ratio per region is the sum of all available feature stage scores divided by the maximum possible score. The maximum possible total stage score is 1.
  The number analyzed represents the number of participants with data at that visit (including imputed values).
Time Frame: Week 24
Population: Full analysis set (All randomized participants who received at least one dose of IP).
Measure: Least Squares Mean (95% Confidence Interval); unit: Grade Score Ratio Change
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 97 | 100
Grade Score Ratio Change | -0.199 [-0.228 to -0.169] | -0.077 [-0.107 to -0.046]
Statistical Analysis 1: Comparison: Benralizumab vs Placebo; Test type: Superiority — For any patients with intercurrent events, the EoE-HSS total stage score after the occurrence of those events were imputed using return-to-baseline MI. Missing data not due to intercurrent events were imputed using MI (MAR); p < 0.0001, ANCOVA; Change from baseline in EoE-HSS TSS = Treatment + baseline EoE-HSS stage score + Region + Baseline steroid use + Presence of strictures at baseline; Difference in Least Squares Means = -0.122, 95% CI 2-sided [-0.16 to -0.09]

6. Secondary Outcome: Changes From Baseline in Centrally-read Endoscopic Reference Score (EREFS)
Description: EREFS is a scoring system for assessing the presence and severity of the major endoscopic signs of EoE.The score ranges from 0 (normal) to 9 (severe disease). EREFS total score (TS): The worst score for each individual component from the proximal and distal scores were summed to form the EREFS total score (TS).
  The number analyzed represents the number of participants with data at that visit (including patients with imputed values post intercurrent events).
Time Frame: Week 24, Week 52
Population: Full analysis set (All randomized participants who received at least one dose of IP).
Measure: Least Squares Mean (95% Confidence Interval); unit: Score
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 85 | 84
Score
  Week 24 | -0.5 [-0.91 to -0.10] | -0.4 [-0.85 to -0.01]
  Week 52: number analyzed (Participants) | 41 | 41
  Week 52 | -0.3 [-0.9 to 0.32] | -0.7 [-1.35 to -0.09]
Statistical Analysis 1: Comparison: Benralizumab vs Placebo; Analysis completed at Week 24; Test type: Superiority — For any patients with intercurrent events, the centrally-read EREFS total score after the occurrence of those events were imputed using return-to-baseline MI. Missing data not due to intercurrent events were imputed using MI (MAR); p = 0.7322, ANCOVA; Model: Change from baseline in EREFS TS = Treatment + baseline EREFS TS + Region + Baseline steroid use + Presence of strictures at baseline; Difference in Least Squares Means = -0.1, 95% CI 2-sided [-0.52 to 0.32]

7. Secondary Outcome: Treatment Responder Rate at Week 24, Defined as a Composite of Histological Response (≤6eos/Hpf) and Clinically Meaningful Improvement From Baseline in Dysphagia Symptom Questionnaire (DSQ) (30% Improvement) at Week 24
Description: Percentage of participants with a treatment response at Week 24. A treatment response is defined as composite of histologic response and clinically meaningful improvement (30% reduction) from baseline in DSQ score. Participants with missing data at Week 24 or with intercurrent events prior to Week 24 are considered non-responders.
Time Frame: Week 24
Population: Full analysis set (All randomized participants who received at least one dose of IP).
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 103 | 107
Percentage of Participants | 43.7 [34.11 to 53.27] | 4.7 [0.67 to 8.67]
Statistical Analysis 1: Comparison: Benralizumab vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 15.86, 95% CI 2-sided [5.79 to 43.47] — Controlling for region (North America and Rest of the world), baseline steroid use, and presence of strictures at baseline. OR values >1 would favor Benra 30 mg treatment group

8. Secondary Outcome: Centrally-read Biopsies for Additional Histopathology Including Tissue Eosinophil Counts at Week 24
Description: Esophagogastroduodenoscopy biopsies were collected at week 24 and sent to the central lab for slide preparation and for central, blinded pathology review of tissue eosinophil counts and histopathology. Centralized slide assessments and scoring from an independent physician review was performed for all biopsies.
Time Frame: Week 24
Population: Full analysis set (All randomized participants who received at least one dose of IP).
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 103 | 107
Participants
  <1 eos/hpf | 84 | 0
  1 to <=6 eos/hpf | 6 | 7
  7 to <15 eos/hpf | 2 | 3
  15 to <60 eos/hpf | 0 | 33
  >=60 eos/hpf | 2 | 56

9. Secondary Outcome: Dysphagia-free Days as Captured by the Dysphagia Symptom Questionnaire (DSQ)
Description: Dysphagia free days is a count ranging from 0-28. Higher counts indicate better outcomes.
  The number analyzed represents the number of participants with data at that visit.
Time Frame: Week 24, Week 52
Population: Full analysis set (All randomized participants who received at least one dose of IP).
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 103 | 107
Days
  Week 24: number analyzed (Participants) | 89 | 93
  Week 24 | 12.65 (10.589) | 16.32 (11.286)
  Week 52: number analyzed (Participants) | 31 | 41
  Week 52 | 19.33 (10.950) | 20.80 (10.472)

10. Secondary Outcome: Frequency of Dysphagia Episodes as Captured by the Eosinophilic Esophagitis Daily Dysphagia Diary (EoE-3D)
Description: EoE-3D is a daily diary focused on the patient experience of EoE. Dysphagia episode frequency is summarized as the total number of dysphagia episodes occurring over each 28-day period following randomization, scaled up to 28 days based on missing days. Requires at least 8 days of evaluable data in each 14-day period within each 28-day period; otherwise the period is set to missing.
  The number analyzed represents the number of participants with data at that visit.
Time Frame: Week 24, Week 52
Population: Full analysis set (All randomized participants who received at least one dose of IP).
Measure: Mean (Standard Deviation); unit: Ratio of Episodes per 28 Day period
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 103 | 107
Ratio of Episodes per 28 Day period
  Week 24: number analyzed (Participants) | 89 | 94
  Week 24 | 20.3 (28.05) | 13.8 (19.15)
  Week 52: number analyzed (Participants) | 31 | 41
  Week 52 | 6.8 (11.59) | 6.2 (9.83)

11. Secondary Outcome: Changes From Baseline in Dysphagia Associated Pain, Discomfort, and Overall Severity as Captured by the Eosinophilic Esophagitis Daily Dysphagia Diary (EoE-3D) at Week 24
Description: In the Eosinophilic Esophagitis Daily Dysphagia Diary (EoE-3D), patients report on whether they experienced episodes of difficulty swallowing in the past 24 hours and if so, how many. Patients respond to 3 questions on the pain, discomfort, and overall severity of the event using a numeric rating scale (0 [no] to 10 [worst]). This is repeated for each episode reported. Each category score is calculated as the sum of daily average values in the 14-day period divided by the number of days with available episodes of difficulty swallowing episodes during the same 14-day period (each of the three final scores range from 0 to 10, with higher values indicating a worse outcome in that category). Requires at least 8 days of evaluable data during the period; otherwise, the mean scores are set to missing. Days with 0 episodes of difficulty swallowing count as evaluable. In case all 14 days with 0 episode of difficulty swallowing, the score is set to missing.
Time Frame: Week 24
Population: Full analysis set (All randomized participants who received at least one dose of IP).
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores per day
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 103 | 107
Scores per day
  Dysphagia-related pain: number analyzed (Participants) | 84 | 73
  Dysphagia-related pain | -0.452 [-0.86 to -0.05] | -0.412 [-0.84 to 0.02]
  Dysphagia-related discomfort: number analyzed (Participants) | 84 | 73
  Dysphagia-related discomfort | -0.370 [-0.73 to -0.01] | -0.189 [-0.57 to 0.19]
  Overall episode severity: number analyzed (Participants) | 84 | 73
  Overall episode severity | -0.481 [-0.83 to -0.13] | -0.137 [-0.51 to 0.24]
Statistical Analysis 1: Comparison: Benralizumab vs Placebo; Dysphagia-related pain; Test type: Superiority — For any patients with intercurrent events, the EoE-3D scores after the occurrence of those events were imputed using return-to-baseline MI. Missing data not due to intercurrent events were imputed using MI (MAR); p = 0.8656, ANCOVA; Model: Change from baseline item score = Treatment + baseline item score + Region + Baseline steroid use + Presence of strictures at baseline; Difference in Least Squares Means = -0.040, 95% CI 2-sided [-0.50 to 0.42]
Statistical Analysis 2: Comparison: Benralizumab vs Placebo; Dysphagia-related discomfort; Test type: Superiority — [test comment as in outcome 11, analysis 1]; p = 0.3926, ANCOVA; [statistical method as in outcome 11, analysis 1]; Difference in Least Squares Means = -0.181, 95% CI 2-sided [-0.60 to 0.23]
Statistical Analysis 3: Comparison: Benralizumab vs Placebo; Overall episode severity; Test type: Superiority — [test comment as in outcome 11, analysis 1]; p = 0.0867, ANCOVA; [statistical method as in outcome 11, analysis 1]; Difference in Least Squares Means = -0.344, 95% CI 2-sided [-0.74 to 0.05]

12. Secondary Outcome: Changes From Baseline in Dysphagia Associated Pain, Discomfort, and Overall Severity as Captured by the Eosinophilic Esophagitis Daily Dysphagia Diary (EoE-3D) at Week 52
Description: as for outcome 11
Time Frame: Week 52
Population: Full analysis set (All randomized participants who received at least one dose of IP).
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores per day
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 46 | 49
Scores per day
  Dysphagia-related pain: number analyzed (Participants) | 24 | 24
  Dysphagia-related pain | -0.511 [-1.40 to 0.38] | -0.776 [-1.65 to 0.10]
  Dysphagia-related discomfort: number analyzed (Participants) | 24 | 24
  Dysphagia-related discomfort | -0.456 [-1.14 to 0.22] | -0.625 [-1.30 to 0.05]
  Overall episode severity: number analyzed (Participants) | 24 | 24
  Overall episode severity | -0.522 [-1.26 to 0.22] | -0.732 [-1.48 to 0.02]

13. Secondary Outcome: Changes From Baseline in Abdominal Pain and Nausea as Captured by the Daily Diary at Week 24
Description: In the Eosinophilic Esophagitis Daily Dysphagia Diary (EoE-3D), respondents are asked to report the severity of abdominal pain and the severity of nausea at their worst over the past 24 hours using an 11-point numeric rating scale (0 [no] to 10 [worst]). Abdominal pain severity and nausea severity will be summarized individually as 14-day mean scores. Each 14-day mean score will be calculated as the sum of daily numerical rating scale score responses divided by the number of days with evaluable data in the same 14-day period. Calculation of the 14-day means will require at least 8 out of 14 days of evaluable data; otherwise, the mean score will be set to missing.
  The number analyzed represents the number of participants with data at that visit (including participants with imputed values post intercurrent events).
Time Frame: Week 24
Population: Full analysis set (All randomized participants who received at least one dose of IP).
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores per day
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 103 | 107
Scores per day
  Abdominal pain severity: number analyzed (Participants) | 95 | 101
  Abdominal pain severity | -0.549 [-0.94 to -0.16] | -0.815 [-1.20 to -0.53]
  Nausea severity: number analyzed (Participants) | 95 | 101
  Nausea severity | -0.524 [-0.90 to -0.15] | -0.820 [-1.19 to -0.45]
Statistical Analysis 1: Comparison: Benralizumab vs Placebo; Abdominal pain severity; Test type: Superiority — [test comment as in outcome 11, analysis 1]; p = 0.2248, ANCOVA; [statistical method as in outcome 11, analysis 1]; Difference in Least Squares Means = 0.267, 95% CI 2-sided [-0.16 to 0.70]
Statistical Analysis 2: Comparison: Benralizumab vs Placebo; Nausea severity; Test type: Superiority — [test comment as in outcome 11, analysis 1]; p = 0.1575, ANCOVA; [statistical method as in outcome 11, analysis 1]; Difference in Least Squares Means = 0.296, 95% CI 2-sided [-0.11 to 0.71]

14. Secondary Outcome: Changes From Baseline in Abdominal Pain and Nausea as Captured by the Daily Diary at Week 52
Description: as for outcome 13
Time Frame: Week 52
Population: Full analysis set (All randomized participants who received at least one dose of IP).
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores per day
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 46 | 49
Scores per day
  Abdominal pain severity: number analyzed (Participants) | 41 | 45
  Abdominal pain severity | -0.826 [-1.44 to -0.22] | -1.039 [-1.62 to -0.46]
  Nausea severity: number analyzed (Participants) | 41 | 45
  Nausea severity | -0.855 [-1.43 to -0.28] | -0.960 [-1.50 to -0.42]

15. Secondary Outcome: Changes From Baseline in the Pediatric Eosinophilic Esophagitis Symptom Severity Module (PEESS)
Description: The Pediatric Eosinophilic Esophagitis Symptom Severity Module, Version 2, Children and Teens Report (PEESS) is an 18-item assessment of EoE symptom severity and frequency validated for use in patients age 8 to 18 years. The recall period is one month. The first 18 questions alternate between a question about a given symptom's frequency (never=0, almost never=1, sometimes=2, often=3, almost always=4) and a question about the symptom's severity (face rating scale with drawings representing: not bad at all=0, a little bad=1, kind of bad=2, bad=3, very bad=4). The remaining two questions ask about frequency of eating less food than others and frequency of needing more time to eat than others. The overall score ranges from 0 to 80, with higher scores representing more severe and frequent EoE symptoms.
  The number analyzed represents the number of participants with data at that visit.
Time Frame: Week 24, Week 52
Population: Full analysis set (All randomized participants who received at least one dose of IP).
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 12 | 9
Score
  Week 24 | -0.8 (11.69) | -5.9 (14.24)
  Week 52: number analyzed (Participants) | 6 | 6
  Week 52 | -6.5 (18.04) | -12.5 (15.67)

16. Secondary Outcome: Changes From Baseline in Adult Eosinophilic Esophagitis Quality of Life Questionnaire (EOE-QoL-A) at Week 24
Description: The Adult Eosinophilic Esophagitis Quality of Life Questionnaire (EoE-QoL-A) is a 30-item assessment developed specifically to measure health-related quality of life in patients with EoE. Responses are on a 5-point scale: Not at all = 4, Slightly = 3, Moderately = 2, Quite a Bit = 1, Extremely = 0. The assessment has 5 domains: eating/diet impact, social impact, emotional impact, disease anxiety and swallowing anxiety.
  Domain scores are calculated as follows:
  * Eating/Diet Impact (range 0 to 40): sum of Q2, Q9, Q16, Q24, Q25, Q26, Q27, Q28, Q29, Q30
  * Social Impact (range 0 to 16): sum of Q14, Q17, Q19, Q22
  * Emotional Impact (range 0 to 32): sum of Q1, Q5, Q6, Q7, Q11, Q13, Q21, Q23
  * Disease Anxiety (range 0 to 20): sum of Q4, Q10, Q12, Q15, Q18,
  * Swallowing Anxiety (range 0 to 12): sum of Q3, Q8, Q20 The total score (range 0 to 120) is calculated as the sum of all responses. Lower scores indicate a greater degree of impairment. Higher scores indicate a better quality of life.
Time Frame: Week 24
Population: Full analysis set (All randomized participants who received at least one dose of IP).
Measure: Least Squares Mean (95% Confidence Interval); unit: Score
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 103 | 107
Score
  Eating/Diet Impact: number analyzed (Participants) | 96 | 96
  Eating/Diet Impact | 1.370 [-0.27 to 3.01] | 1.169 [-0.46 to 2.79]
  Social Impact: number analyzed (Participants) | 96 | 96
  Social Impact | 1.095 [0.21 to 1.98] | 0.948 [0.07 to 1.83]
  Emotional Impact: number analyzed (Participants) | 96 | 96
  Emotional Impact | 0.912 [-0.46 to 2.29] | 0.902 [-0.46 to 2.27]
  Disease Anxiety: number analyzed (Participants) | 96 | 96
  Disease Anxiety | 0.185 [-0.77 to 1.14] | -0.201 [-1.15 to 0.75]
  Swallowing Anxiety: number analyzed (Participants) | 96 | 96
  Swallowing Anxiety | 0.443 [-0.23 to 1.12] | 0.605 [-0.06 to 1.27]
  Total Score: number analyzed (Participants) | 96 | 96
  Total Score | 4.380 [-0.36 to 9.12] | 3.362 [-1.33 to 8.06]
Statistical Analysis 1: Comparison: Benralizumab vs Placebo; Eating/Diet Impact; Test type: Superiority — For any patients with intercurrent events, the EoE-QoL-A scores after the occurrence of those events were imputed using return-to-baseline MI. Missing data not due to intercurrent events were imputed using MI (MAR); p = 0.8239, ANCOVA; [statistical method as in outcome 11, analysis 1]; Difference in Least Squares Means = 0.202, 95% CI 2-sided [-1.57 to 1.98]
Statistical Analysis 2: Comparison: Benralizumab vs Placebo; Social Impact; Test type: Superiority — [test comment as in outcome 16, analysis 1]; p = 0.7623, ANCOVA; [statistical method as in outcome 11, analysis 1]; Difference in Least Squares Means = 0.147, 95% CI 2-sided [-0.80 to 1.10]
Statistical Analysis 3: Comparison: Benralizumab vs Placebo; Emotional Impact; Test type: Superiority — [test comment as in outcome 16, analysis 1]; p = 0.9898, ANCOVA; [statistical method as in outcome 11, analysis 1]; Difference of Least Squares Means = 0.010, 95% CI 2-sided [-1.47 to 1.49]
Statistical Analysis 4: Comparison: Benralizumab vs Placebo; Disease Anxiety; Test type: Superiority — [test comment as in outcome 16, analysis 1]; p = 0.4603, ANCOVA; [statistical method as in outcome 11, analysis 1]; Difference in Least Squares Means = 0.386, 95% CI 2-sided [-0.64 to 1.41]
Statistical Analysis 5: Comparison: Benralizumab vs Placebo; Swallowing Anxiety; Test type: Superiority — [test comment as in outcome 16, analysis 1]; p = 0.6613, ANCOVA; [statistical method as in outcome 11, analysis 1]; Difference in Least Squares Means = -0.162, 95% CI 2-sided [-0.89 to 0.56]
Statistical Analysis 6: Comparison: Benralizumab vs Placebo; Total Score; Test type: Superiority — [test comment as in outcome 16, analysis 1]; p = 0.6965, ANCOVA; [statistical method as in outcome 11, analysis 1]; Difference in Least Squares Means = 1.017, 95% CI 2-sided [-4.09 to 6.13]

17. Secondary Outcome: Changes From Baseline in Adult Eosinophilic Esophagitis Quality of Life Questionnaire (EOE-QoL-A) at Week 52
Description: as for outcome 16
Time Frame: Week 52
Population: Full analysis set (All randomized participants who received at least one dose of IP).
Measure: Least Squares Mean (95% Confidence Interval); unit: Score
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 46 | 48
Score
  Eating/Diet Impact: number analyzed (Participants) | 43 | 47
  Eating/Diet Impact | 1.408 [-1.01 to 3.83] | 1.949 [-0.32 to 4.21]
  Social Impact: number analyzed (Participants) | 43 | 47
  Social Impact | 1.462 [0.09 to 2.83] | 1.984 [0.70 to 3.27]
  Emotional Impact: number analyzed (Participants) | 43 | 47
  Emotional Impact | 1.768 [-0.21 to 3.75] | 2.451 [0.58 to 4.33]
  Disease Anxiety: number analyzed (Participants) | 43 | 47
  Disease Anxiety | 1.063 [-0.43 to 2.56] | 1.152 [-0.27 to 2.57]
  Swallowing Anxiety: number analyzed (Participants) | 43 | 47
  Swallowing Anxiety | 0.677 [-0.37 to 1.72] | 1.085 [0.10 to 2.07]
  Total Score: number analyzed (Participants) | 43 | 47
  Total Score | 6.749 [-0.35 to 13.84] | 8.714 [2.03 to 15.40]

18. Secondary Outcome: Change From Baseline in Short Form 36-item Health Survey (Version 2, Acute Recall) (SF-36v2) at Week 24
Description: The Short Form 36-item Health Survey, version 2, acute recall (SF-36v2) is a 36-item, self-report survey of functional health and well-being, with a 1-week recall period. There are 8 domain scores: Physical Functioning (PF), Role Limitations due to Physical Health (RP), Bodily Pain (BP), General Health Perceptions (GH), Vitality (VT), Social Functioning (SF), Role Limitations due to Emotional Problems (RE), and Mental Health (MH). Psychometrically-based physical and mental health component summary scores (PCS and MCS, respectively) were computed from subscale scores to give a broader metric of physical and mental health-related quality of life. All scores range from 0-100, with higher scores meaning better outcomes.
  The number analyzed represents the number of participants with data at that visit (including participants with imputed values post intercurrent events).
Time Frame: Week 24
Population: Full analysis set (All randomized participants who received at least one dose of IP).
Measure: Least Squares Mean (95% Confidence Interval); unit: Score
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 83 | 81
Score
  Physical functioning (PF) | 0.2 [-1.36 to 1.70] | 0.5 [-0.98 to 1.97]
  Role limitations due to physical health (RP) | 0.5 [-1.03 to 2.10] | 1.5 [-0.06 to 2.99]
  Bodily pain (BP) | -0.6 [-2.92 to 1.82] | 0.2 [-2.07 to 2.53]
  General health perceptions (GH) | -0.9 [-2.62 to 0.78] | -0.9 [-2.54 to 0.76]
  Vitality (VT) | -0.5 [-2.47 to 1.54] | -0.5 [-2.50 to 1.48]
  Social functioning (SF) | -1.5 [-3.84 to 0.92] | 0.1 [-2.26 to 2.39]
  Role limitations due to emotional problems (RE) | -1.1 [-3.68 to 1.51] | -0.4 [-2.95 to 2.15]
  Mental health (MH) | -1.7 [-3.83 to 0.51] | -0.8 [-2.91 to 1.31]
  Psychometrically-based physical summary score (PCS) | 0.4 [-1.21 to 2.01] | 0.8 [-0.75 to 2.34]
  Mental health component summary scores (MCS) | -1.8 [-4.10 to 0.53] | -1.2 [-3.44 to 1.11]
Statistical Analysis 1: Comparison: Benralizumab vs Placebo; Physical functioning (PF); Test type: Superiority — For any patients with intercurrent events, the SF-36 domain scores after the occurrence of those events were imputed using return-to-baseline MI. Missing data not due to intercurrent events were imputed using MI (MAR); p = 0.6852, ANCOVA; [statistical method as in outcome 11, analysis 1]; Difference in Least Squares Means = -0.3, 95% CI 2-sided [-1.93 to 1.27]
Statistical Analysis 2: Comparison: Benralizumab vs Placebo; Role limitations due to physical health (RP); Test type: Superiority — [test comment as in outcome 18, analysis 1]; p = 0.2685, ANCOVA; [statistical method as in outcome 11, analysis 1]; Difference in Least Squares Means = -0.9, 95% CI 2-sided [-2.57 to 0.72]
Statistical Analysis 3: Comparison: Benralizumab vs Placebo; Bodily pain (BP); Test type: Superiority — [test comment as in outcome 18, analysis 1]; p = 0.5380, ANCOVA; [statistical method as in outcome 11, analysis 1]; Difference in Least Squares Means = -0.8, 95% CI 2-sided [-3.27 to 1.71]
Statistical Analysis 4: Comparison: Benralizumab vs Placebo; General health perceptions (GH); Test type: Superiority — [test comment as in outcome 18, analysis 1]; p = 0.9734, ANCOVA; [statistical method as in outcome 11, analysis 1]; Difference in Least Squares Means = -0.0, 95% CI 2-sided [-1.81 to 1.75]
Statistical Analysis 5: Comparison: Benralizumab vs Placebo; Vitality (VT); Test type: Superiority — [test comment as in outcome 18, analysis 1]; p = 0.9653, ANCOVA; [statistical method as in outcome 11, analysis 1]; Difference in Least Squares Means = 0.0, 95% CI 2-sided [-2.09 to 2.19]
Statistical Analysis 6: Comparison: Benralizumab vs Placebo; Social functioning (SF); Test type: Superiority — [test comment as in outcome 18, analysis 1]; p = 0.2326, ANCOVA; [statistical method as in outcome 11, analysis 1]; Difference in Least Squares Means = -1.5, 95% CI 2-sided [-4.04 to 0.98]
Statistical Analysis 7: Comparison: Benralizumab vs Placebo; Role limitations due to emotional problems (RE); Test type: Superiority — [test comment as in outcome 18, analysis 1]; p = 0.6274, ANCOVA; [statistical method as in outcome 11, analysis 1]; Difference in Least Squares Means = -0.7, 95% CI 2-sided [-3.44 to 2.08]
Statistical Analysis 8: Comparison: Benralizumab vs Placebo; Mental health (MH); Test type: Superiority — [test comment as in outcome 18, analysis 1]; p = 0.4599, ANCOVA; [statistical method as in outcome 11, analysis 1]; Difference in Least Squares Means = -0.9, 95% CI 2-sided [-3.14 to 1.42]
Statistical Analysis 9: Comparison: Benralizumab vs Placebo; Psychometrically-based physical summary score (PCS); Test type: Superiority — [test comment as in outcome 18, analysis 1]; p = 0.6456, ANCOVA; [statistical method as in outcome 11, analysis 1]; Difference in Least Squares Means = -0.4, 95% CI 2-sided [-2.07 to 1.28]
Statistical Analysis 10: Comparison: Benralizumab vs Placebo; Mental health component summary scores (MCS); Test type: Superiority — [test comment as in outcome 18, analysis 1]; p = 0.6206, ANCOVA; [statistical method as in outcome 11, analysis 1]; Difference in Least Squares Means = -0.6, 95% CI 2-sided [-3.08 to 1.84]

19. Secondary Outcome: Change From Baseline in Short Form 36-item Health Survey (Version 2, Acute Recall) (SF-36v2) at Week 52
Description: as for outcome 18
Time Frame: Week 52
Population: Full analysis set (All randomized participants who received at least one dose of IP).
Measure: Least Squares Mean (95% Confidence Interval); unit: Score
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 46 | 48
Score
  Physical functioning (PF): number analyzed (Participants) | 34 | 38
  Physical functioning (PF) | 0.3 [-1.86 to 2.51] | 0.4 [-1.60 to 2.46]
  Role limitations due to physical health (RP): number analyzed (Participants) | 34 | 38
  Role limitations due to physical health (RP) | -0.5 [-3.27 to 2.20] | 0.9 [-1.63 to 3.51]
  Bodily pain (BP): number analyzed (Participants) | 34 | 38
  Bodily pain (BP) | 0.6 [-2.69 to 3.97] | 1.8 [-1.34 to 5.00]
  General health perceptions (GH): number analyzed (Participants) | 34 | 38
  General health perceptions (GH) | 2.3 [-0.71 to 5.39] | 0.7 [-2.17 to 3.59]
  Vitality (VT): number analyzed (Participants) | 34 | 38
  Vitality (VT) | -0.2 [-2.69 to 2.31] | -2.0 [-4.42 to 0.44]
  Social functioning (SF): number analyzed (Participants) | 34 | 38
  Social functioning (SF) | 0.2 [-3.73 to 4.17] | -0.5 [-4.26 to 3.34]
  Role limitations due to emotional problems (RE): number analyzed (Participants) | 34 | 38
  Role limitations due to emotional problems (RE) | -0.1 [-3.30 to 3.19] | -0.3 [-3.39 to 2.76]
  Mental health (MH): number analyzed (Participants) | 34 | 38
  Mental health (MH) | 1.2 [-1.37 to 3.69] | -1.1 [-3.46 to 1.30]
  Psychometrically-based physical summary score (PCS): number analyzed (Participants) | 34 | 38
  Psychometrically-based physical summary score (PCS) | 0.5 [-2.15 to 3.18] | 1.4 [-1.15 to 3.85]
  Mental health component summary scores (MCS): number analyzed (Participants) | 34 | 38
  Mental health component summary scores (MCS) | 0.5 [-2.44 to 3.50] | -1.9 [-4.78 to 0.89]

20. Secondary Outcome: Percent of Patients With Relevant Concomitant Procedures and Healthcare Resource Utilization at Week 24 and Week 52.
Description: Percent of patients with any relevant concomitant procedures or healthcare resource utilization for Eosinophilic esophagitis (EoE) or an EoE-related episode (e.g., an intervention for food impaction or stricture requiring dilatation) since last healthcare resource utilization assessment during the previous scheduled visit. Assessed at Week 24 and Week 52.
Time Frame: Week 24, Week 52
Population: Full analysis set (All randomized participants who received at least one dose of IP).
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 103 | 107
Participants
  Week 24 | 3 | 5
  Week 52 | 0 | 2

21. Secondary Outcome: Patient Reported Overall Severity of Disease as Measured by Patient Global Impression of Severity (PGI-S) at Week 24
Description: Patient Global Impression of Severity (PGI-S) is an assessment of the patient's perceived disease severity. The answer options are "no symptoms," "very mild," "mild," "moderate," "severe," and "very severe."
  The number analyzed represents the participants with evaluable PGI-S results at that timepoint.
Time Frame: Week 24
Population: Full analysis set (All randomized participants who received at least one dose of IP).
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 96 | 95
Participants
  No symptoms | 4 | 11
  Very mild | 23 | 27
  Mild | 34 | 32
  Moderate | 29 | 17
  Severe | 3 | 6
  Very Severe | 3 | 2

22. Secondary Outcome: Patient Reported Overall Severity of Disease as Measured by Patient Global Impression of Severity (PGI-S) at Week 52
Description: as for outcome 21
Time Frame: Week 52
Population: Full analysis set (All randomized participants who received at least one dose of IP).
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 36 | 42
Participants
  No symptoms | 6 | 10
  Very mild | 12 | 14
  Mild | 9 | 13
  Moderate | 8 | 5
  Severe | 0 | 0
  Very Severe | 1 | 0

23. Secondary Outcome: Patient Reported Change in Health Status Since Baseline as Measured by Patient Global Impression of Change (PGI-C) at Week 24
Description: Patient Global Impression of Change (PGI-C) measures the patient's overall impression of response to treatment since the initial dose. The answer options are "much better," "moderately better," "a little better," "about the same/no change," "a little worse," "moderately worse," and "much worse."
  The number analyzed represents the participants with evaluable PGI-C results at that timepoint.
Time Frame: Week 24
Population: Full analysis set (All randomized participants who received at least one dose of IP).
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 96 | 96
Participants
  Much better | 13 | 13
  Moderately better | 13 | 17
  A little better | 21 | 20
  About the same | 37 | 36
  A little worse | 7 | 6
  Moderately worse | 3 | 3
  Much worse | 2 | 1

24. Secondary Outcome: Patient Reported Change in Health Status Since Baseline as Measured by Patient Global Impression of Change (PGI-C) at Week 52
Description: as for outcome 23
Time Frame: Week 52
Population: Full analysis set (All randomized participants who received at least one dose of IP).
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 36 | 43
Participants
  Much better | 12 | 13
  Moderately better | 3 | 12
  A little better | 8 | 12
  About the same | 9 | 6
  A little worse | 4 | 0
  Moderately worse | 0 | 0
  Much worse | 0 | 0

25. Other Pre Specified Outcome: Benralizumab Pharmacokinetics
Description: Serum concentrations of benralizumab through Week 52. Geometric mean calculated using log transformed data.
Time Frame: Up to week 52
Population: PK analysis set (All participants who received benralizumab and who had at least one quantifiable serum PK observation post first dose).
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 97 | 96
ng/mL
  Week 8: number analyzed (Participants) | 95 | 0
  Week 8 | 1555.70 [1425.31 to 1698.02] |
  Week 16: number analyzed (Participants) | 91 | 0
  Week 16 | 1582.46 [1322.66 to 1893.30] |
  Week 24: number analyzed (Participants) | 85 | 91
  Week 24 | 1338.65 [1027.05 to 1744.78] | NA [NA to NA] — Below limit of quantification
  Week 36: number analyzed (Participants) | 67 | 63
  Week 36 | 1405.94 [985.94 to 2004.86] | 1362.27 [1051.69 to 1764.58]
  Week 52: number analyzed (Participants) | 30 | 36
  Week 52 | 1278.13 [749.19 to 2180.52] | 1495.61 [975.73 to 2292.50]

26. Other Pre Specified Outcome: Immunogenicity of Benralizumab in Double Blind Period
Description: Immunogenicity of benralizumab assessed by ADA and nAb in the Double Blind period.
Time Frame: Up to Week 24
Population: Safety analysis set (All participants who received at least one dose of IP).
Measure: Number; unit: Participants
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 103 | 107
Participants
  ADA positive/ADA prevalence (positive at baseline and/or post-baseline) | 18 | 8
  ADA negative (negative at all assessments) | 85 | 99
  Treatment-emergent ADA positive/ADA incidence: number analyzed (Participants) | 102 | 106
  Treatment-emergent ADA positive/ADA incidence | 18 | 4
  ADA persistently positive: number analyzed (Participants) | 102 | 106
  ADA persistently positive | 18 | 3
  ADA positive subjects with maximum titre > median of maximum titres | 6 | 4
  nAb positive/nAb prevalence | 10 | 0
  ADA persistently positive and nAb positive: number analyzed (Participants) | 102 | 107
  ADA persistently positive and nAb positive | 10 | 0

27. Other Pre Specified Outcome: Immunogenicity of Benralizumab in Double Blind + Open Label Periods
Description: Immunogenicity of benralizumab assessed by ADA and nAb in the Double Blind and Open Label periods.
Time Frame: Up to Week 52
Population: Safety analysis set (All participants who received at least one dose of IP).
Measure: Number; unit: Participants
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 103 | 107
Participants
  ADA positive/ADA prevalence (positive at baseline and/or post-baseline): number analyzed (Participants) | 103 | 105
  ADA positive/ADA prevalence (positive at baseline and/or post-baseline) | 19 | 17
  ADA negative (negative at all assessments): number analyzed (Participants) | 103 | 105
  ADA negative (negative at all assessments) | 84 | 88
  Treatment-emergent ADA positive/ADA incidence: number analyzed (Participants) | 102 | 105
  Treatment-emergent ADA positive/ADA incidence | 19 | 11
  ADA persistently positive: number analyzed (Participants) | 102 | 105
  ADA persistently positive | 16 | 10
  ADA positive subjects with maximum titre > median of maximum titres: number analyzed (Participants) | 103 | 105
  ADA positive subjects with maximum titre > median of maximum titres | 7 | 7
  nAb positive/nAb prevalence: number analyzed (Participants) | 103 | 105
  nAb positive/nAb prevalence | 10 | 5
  ADA persistently positive and nAb positive: number analyzed (Participants) | 102 | 105
  ADA persistently positive and nAb positive | 10 | 5

28. Other Pre Specified Outcome: Safety and Tolerability in Double Blind Period
Description: Percentage of participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) in the Double Blind treatment period (up to Week 24).
Time Frame: Up to Week 24
Population: Safety analysis set (All participants who received at least one dose of IP).
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 103 | 107
Participants
  Any AE | 66 | 66
  Any SAE | 2 | 1

29. Other Pre Specified Outcome: Safety and Tolerability in the Open Label Period
Description: Percentage of participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) in the Open Label treatment period (past week 24).
Time Frame: From Week 24 up to Week 52
Population: Safety analysis set (All participants who received at least one dose of IP).
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 100 | 105
Participants
  Any AE | 53 | 60
  Any SAE | 2 | 4

ADVERSE EVENTS:
Time Frame: On study AEs were collected from the first dose to the last date in study, up to 104 weeks.
Description: Benra 30 mg = all participants who initially received Benralizumab in the double-blind (DB) period and continued to receive Benralizumab in the open-label (OL) and open-label extension (OLE) period. Placebo = all participants who initially received Placebo in the DB period, up to week 24. All Benra = all participants who initially received Benralizumab in the DB period + all participants who received Benralizumab in the OL and OLE periods.
Groups:
- Benra 30 mg: 30mg Benralizumab injection delivered subcutaneously every 4 weeks
- Placebo: Matching Placebo injection delivered subcutaneously every 4 weeks through week 24
- All Benra: Participants who were received 30 mg Benralizumab injection delivered every 4 weeks during double-blind period, up to week 24 + participants who received 30 mg Benralizumab injection delivered every 4 weeks during the open-label and open-label extension periods, after week 24 (i.e. all participants who received Benra in any period).
Arm/Group | Benra 30 mg | Placebo | All Benra
All-Cause Mortality (participants affected / at risk) | 0/103 | 0/107 | 0/208
Serious Adverse Events (participants affected / at risk) | 4/103 | 1/107 | 9/208
Other Adverse Events (participants affected / at risk) | 60/103 | 42/107 | 95/208
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benra 30 mg (N=103) | Placebo (N=107) | All Benra (N=208)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Affective disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Disruptive mood dysregulation disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Oppositional defiant disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (2) | 0 (0) | 1 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oesophageal food impaction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)
Oesophageal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benra 30 mg (N=103) | Placebo (N=107) | All Benra (N=208)
Nasopharyngitis (Infections and infestations) | 12 (20) | 6 (6) | 19 (29)
Pharyngitis (Infections and infestations) | 5 (5) | 0 (0) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 5 (6) | 8 (9)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 4 (4) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 6 (7)
Headache (Nervous system disorders) | 12 (15) | 11 (16) | 14 (18)
Asthma (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4) | 9 (10)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 3 (4) | 11 (14)
Hypertension (Vascular disorders) | 4 (4) | 0 (0) | 5 (5)
Nausea (Gastrointestinal disorders) | 4 (4) | 3 (3) | 5 (5)
Injection site erythema (General disorders) | 5 (13) | 2 (2) | 7 (15)
Pyrexia (General disorders) | 3 (3) | 1 (2) | 7 (7)
Immunisation reaction (Immune system disorders) | 4 (4) | 1 (1) | 4 (4)
COVID-19 (Infections and infestations) | 34 (38) | 13 (13) | 49 (53)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Institution and/or the Principal Investigator shall not include in or shall remove from any proposed publication any Confidential Information, errors or inaccuracies; and shall withhold publication, submission for publication or presentation for a period of ninety (90) days from the date on which the Company receives the material to allow the Company to take such measures as the Company considers necessary to preserve its proprietary rights and/or protect its Confidential Information.

DOCUMENTS (2):
  • Study Protocol (2022-04-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT04543409/Prot_004.pdf
  • Statistical Analysis Plan (2022-09-02): https://cdn.clinicaltrials.gov/large-docs/09/NCT04543409/SAP_005.pdf